CLINICAL TRIAL: NCT06326398
Title: The Effect of Using 3D Printers and Moulage on Improving Stoma Care Knowledge and Skills in Nursing Students
Brief Title: The Effect of Using 3D Printers and Moulage on Improving Stoma Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Tülin YILDIZ, Prof. Dr., Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3D moulage
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Stoma Colostomy
Keywords: stoma; nursing student; 3d printer; moulage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will perform stoma care using the low-reality simulation (stoma model) method.
- Experimental group (Experimental): Students in the experimental group will perform stoma care using high-reality simulation (3D printing and moulage) method.
  Interventions: Other: Stoma Care

INTERVENTIONS:
Other: Stoma Care — Nursing students practice stoma care with low and high fidelity simulation
  Arms: Experimental group

SUMMARY:
When studies in the literature are examined, there are studies in which various methods are applied to students' stoma care knowledge and skills. Additionally, it is seen that there are studies using moulage or 3D printers as simulation applications in nursing education. However, there is no study on high-reality simulation application using 3D printer and moulage technique together.nIn this research, the effect of the stoma created with a 3D printer in a high-reality simulation on the stoma care knowledge and skills, satisfaction and self-confidence of nursing students will be examined by using the moulage technique. In addition, this application will be compared with nursing students' stoma care practices in the stoma model, which is classified as low-reality simulation. We think that our project will be unique in this field, as it uses current technological methods together in this planned research and is different from similar studies.

DETAILED DESCRIPTION:
A stoma is an opening created by inserting an organ into the skin using a surgical method. Colostomy, ileostomy and urostomy, in which excretion is provided through an opening created on the anterior wall of the abdomen outside normal anatomical pathways, are among the most commonly created stomas. Although stomas are created for various reasons, they are most commonly opened due to colorectal and bladder cancers.

According to the International Agency for Research on Cancer (IARC), colorectal cancer ranks 3rd and bladder cancer ranks 10th in all ages and genders. Although the exact number of individuals with a stoma worldwide is unknown, it is estimated that 18-35% of individuals diagnosed with cancer have to live with a stoma temporarily or permanently during the treatment process. In this regard, it is thought that the number of individuals with stoma will increase with the increase in colorectal and bladder cancers. This increase also increases the need for nursing care of individuals with stoma. Accordingly, it is important to provide this care skill to nursing students, who are the nurses of the future, during nursing education.

Nursing education; It includes multifaceted education and training activities including theoretical, laboratory and application areas. It is thought that students who gain sufficient knowledge and experience about stoma care during their studies provide effective care to individuals with stomas when they start working as professional nurses, and that their adaptation to stoma and quality of life increases with this care. Stoma care is among the basic nursing skills that nurses apply autonomously. While training student nurses on stoma care, methods that improve their cognitive, sensory and psychomotor skills should be used. In this context, with technological developments, various methods such as computer systems and simulation applications are becoming widespread in nursing education day by day.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research,
* Not taking the Surgical Diseases Nursing course before,
* Not having received stoma care training before,
* Not having observed stoma care in previous applied courses
* Giving both written and verbal permission to participate in the research

Exclusion Criteria:

* Refusal to participate in the research,
* Receiving training on stoma care,
* Observing or performing stoma care before,
* Having a high school or associate degree related to the field of health

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level Evaluation Form Regarding Stoma Care | Pre-intervention and immediately after the intervention
  Measuring stoma care knowledge
Stoma Care Skill Grading Key | Immediately after the intervention
  This tool consists of 23 items containing stoma care process steps. In the Rubric, the adequacy is scored between 0-2 (0- Insufficient, 1- Partially adequate, 2- Sufficient) for each process step. A minimum of 0 and a maximum of 46 points can be obtained from the Rubric. The total score received from the Rubric indicates the adequacy of stoma care skills.
Student Satisfaction and Self-Confidence Scale in Learning | Immediately after the intervention
  Measuring satisfaction and self-confidence

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ambe PC, Kurz NR, Nitschke C, Odeh SF, Moslein G, Zirngibl H. Intestinal Ostomy. Dtsch Arztebl Int. 2018 Mar 16;115(11):182-187. doi: 10.3238/arztebl.2018.0182. PMID 29607805
- [Background] Bucknall TK, Forbes H, Phillips NM, Hewitt NA, Cooper S, Bogossian F; FIRST2ACT Investigators. An analysis of nursing students' decision-making in teams during simulations of acute patient deterioration. J Adv Nurs. 2016 Oct;72(10):2482-94. doi: 10.1111/jan.13009. Epub 2016 Jun 5. PMID 27265550
- See also: 12. International Agency for Research on Cancer (IARC), 2020. "Cancer Today" — http://gco.iarc.fr/today/home